CLINICAL TRIAL: NCT00094926
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Study of the Effectiveness and Safety of RISPERDAL CONSTA Augmentation in Adult Patients With Frequently-relapsing Bipolar Disorder
Brief Title: A Study of Effectiveness and Safety of Risperdal CONSTA Added to Usual Treatment in Patients With Bipolar Disorder Who Have Frequent Mood Episodes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sr Director, Clinical Development Leader, Ortho McNeil Janssen Scientific Affairs, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR004693; RISBIP302
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Bipolar Disorder
Keywords: Risperidal CONSTA; Bipolar disorder; mood episodes; Safety and efficacy, adjuvant therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 001 (Experimental)
  Interventions: Drug: Risperdal Consta
- 002 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Risperdal Consta — 25, 37.5 or 50mg IM injections every 2wks for 52wks
  Arms: 001
Drug: placebo — matching placebo IM injections every 2wks for 52wks
  Arms: 002

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of the long acting injectable form of the atypical antipsychotic Risperidone (Risperdal CONSTA), along with treatment as usual (TAU), in bipolar disorder patients who had more than 4 mood episodes in the past year.

DETAILED DESCRIPTION:
Frequently-relapsing (more than 4 episodes in the last year) bipolar patients are a sub-group of patients who have multiple mood episodes in spite of treatment. Currently available treatments may have little impact on number and frequency of manic and/or depressed mood episodes and as a result, these patients have higher than average rates of illness and death. This study examines the effectiveness and side effects of risperidone long-acting injections (LAI) added to treatment as usual (TAU) in frequently-relapsing bipolar patients. The study has two main phases. The first phase is open-label (patients and doctors know what medication and dose the patient is receiving- both risperidone LAI and TAU) and lasts 16 weeks. During that time, patients are treated with the goal that they reach "remission", a predefined level of improvement (decrease in number and severity of mood episodes.) Patients who meet remission criteria at the end of the first phase are randomized (like flipping a coin) to either continue receiving the same dose of risperidone LAI plus TAU, or placebo injections plus TAU. Patients continue in the second phase for 52 weeks, during which time the effectiveness is measured by time to "relapse" (worsening of mood symptoms severe enough to require hospitalization or a major change in medication.) Additional effectiveness, safety, and side effect measures are evaluated throughout the length of the study.

Long-acting risperidone injection 25 mg will be administered every two weeks through a gluteal injection for at least one month. Thereafter, the dose may be increased to 37.5mg then to 50 mg based on clinical response and tolerability. Supplemental use of oral Risperdal (1 to 2 mg/day) will be permitted during the first 12 weeks of the Open-Label Stabilization Phase. Patients must be taking a stable dose of risperidone LAI for the 4 weeks immediately prior to entering the Double-Blind Phase.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Must agree to receive regular injections
* Must have current diagnosis of bipolar disorder I or II
* Must have at least four episodes of mood disorder in the last year that required psychiatric intervention

Exclusion Criteria:

* Female who is or may be pregnant or breastfeeding, who is not at least 1 year postmenopausal, or is not using reliable and adequate birth control
* Psychiatric diagnosis is due directly to effects of a substance or general medical condition
* Substance dependence
* Received treatment with a long-acting injectable antipsychotic less than 2 injection cycles prior to baseline (so, for example, if the drug is injected every 2 weeks, the patient could not enroll in the study if they had received an injection within the last 4 weeks)
* Received Electroconvulsive Therapy (ECT) within the last month
* Began psychotherapy ("talk therapy") within 2 months
* In the past month was treated with any of these medications: carbamazepine, oxcarbazepine, fluoxetine, paroxetine, or clozapine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2004-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Efficacy will be determined by measuring the time (in days) from randomization to event/relapse; relapse will be assessed by clinical status, rating scale changes, and pharmacologic stability in double-blind phase. | 52 weeks

SECONDARY OUTCOMES:
Safety and tolerability as assessed by adverse event reports (every 2 weeks), scores on movement disorder measures, laboratory parameters, vital signs, ECG measures and physical examination reports (every 2-3 months) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Macfadden W, Alphs L, Haskins JT, Turner N, Turkoz I, Bossie C, Kujawa M, Mahmoud R. A randomized, double-blind, placebo-controlled study of maintenance treatment with adjunctive risperidone long-acting therapy in patients with bipolar I disorder who relapse frequently. Bipolar Disord. 2009 Dec;11(8):827-39. doi: 10.1111/j.1399-5618.2009.00761.x. PMID 19922552
- See also: Adjunctive Risperdal Consta Study in Frequently Relapsing Bipolar Disorder Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=623&filename=CR004693_CSR.pdf